CLINICAL TRIAL: NCT05799417
Title: Brain Oscillatory Signatures of Auditory Stimuli Across Different Vigilance and Sedation States
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-00970
Record Dates: First submitted 2023-03-01; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia; Sleep

STUDY DESIGN:
Intervention Model Description: The investigators forecast a maximal enrollment of 80 participants. However, an interim-analysis will be conducted after 10-14 participants to check estimated effect-size of intervention.
Masking Description: This study is designed as non-randomized clinical study where acoustic stimuli of different characteristics are played and compared to within-subject baselines across various sedation and/or sleep states.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acoustic stimuli (Experimental): Acoustic stimuli and comparison to within-subject baseline
  Interventions: Other: Acoustic stimuli

INTERVENTIONS:
Other: Acoustic stimuli — During different states of sedation/anaesthesia and sleep, acoustic stimuli will be presented and compared to a within-subject baseline.

SUMMARY:
The investigators want to explore how presenting acoustic stimuli influences brain oscillatory signatures and heart rhythm- dynamics across different vigilance and sedation states.

The investigators will administer acoustic stimuli during sedation and anaesthesia while brain activity and heart activity are being recorded by electroencephalogram and electrocardiogram.

On the day following anaesthesia an optional nap/sleep period's EEG and ECG will be recorded. During this short sleep, patients will again be exposed to acoustic stimuli. The recorded EEG and ECG will be compared intra-and inter-individually to recordings from sedation and anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Good general health status
* Planned ophthalmic/plastic surgery at Inselspital Berne

Exclusion Criteria:

* Contraindications on ethical grounds
* Neurological/neurodegenerative disorder
* Hearing problems (only if patients are not able to perceive the acoustic stimuli)
* Pacemaker
* Deep brain stimulator
* Pregnancy
* Known or suspected drug or alcohol abuse
* Critical surgery procedure

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Brain oscillatory power derived by EEG | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Brain oscillatory response to acoustic stimuli derived by power spectral density in canonical frequency bands from 0.5 up to 40 Hz.
Brain oscillatory response derived by Hilbert Amplitude | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Brain oscillatory response to acoustic stimuli derived by Hilbert-transforming EEG data and extracting Hilbert amplitude in microVolts
Spindle characteristics - number of spindles | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Number of spindles
Spindle characteristics - amplitude of spindles | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Spindle amplitude in microVolts
Spindle characteristics - frequency of spindles | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Frequency of spindles in Hz
Spindle characteristics - duration of spindles | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Duration of spindles in ms

SECONDARY OUTCOMES:
Heart rate | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Heart rate derived from echocardiogram in bpm
Instantaneous heart rate | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Instantaneous heart rate derived from echocardiogram in bpm
Heart rate variability | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Heart rate variability derived from echocardiogram in ms
Slow wave characteristics - amplitude | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Slow wave amplitude in microVolt
Slow wave characteristics - number | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Number of slow waves
Slow wave characteristics - frequency | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Frequency of slow waves in Hz
Slow wave characteristics - slope | Continuously across anaesthesia/sedation/sleep up to 8 hours
  Slope of slow waves in microVolts/s
Number of sleep arousals | Continuously across sleep up to 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Lersch, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No